CLINICAL TRIAL: NCT07200154
Title: A Single-arm、Exploratory Study of Adebrelimab in Combination With Chemoradiotherapy Followed by Adebrelimab Maintenance in Patients With Limited-stage Small-cell Lung Cancer
Brief Title: Adebrelimab Plus Chemoradiotherapy Followed by Adebrelimab Maintenance in Limited-Stage SCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025YJZ78
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Limited-stage Small-cell Lung Cancer; Concurrent Chemoradiation Therapy
Keywords: limited-stage small-cell lung cancer; Immune checkpoint inhibitors; Concurrent Chemoradiation Therapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental group (Experimental): Patients meeting inclusion criteria will receive adebrelimab combined with chemotherapy followed by concurrent radiotherapy. Adebrelimab maintenance therapy will be administered until disease progression or intolerable toxicity, for a maximum duration of 2 years.
  Interventions: Drug: Adebrelimab with concurrent chemoradiotherapy

INTERVENTIONS:
Drug: Adebrelimab with concurrent chemoradiotherapy — Adebrelimab combined with chemotherapy and concurrent radiotherapy, followed by maintenance therapy with Adebrelimab until disease progression or intolerable toxicity, for up to 2 years.

SUMMARY:
This is a single-arm, open-label, single-center phase II trial that will enroll 30 patients with limited-stage small-cell lung cancer to evaluate the safety and efficacy of adebrelimab combined with chemoradiotherapy followed by adebrelimab maintenance.

DETAILED DESCRIPTION:
This investigator-initiated trial will be conducted in the Department of Radiation Oncology, Peking University Cancer Hospital. Thirty patients with limited-stage small-cell lung cancer (LS-SCLC) will be enrolled in this pilot study to explore whether the addition of adebrelimab to chemoradiotherapy can improve outcomes for this population.

Eligible participants will receive adebrelimab combined with chemoradiotherapy（etoposide plus platinum). Patients who achieve complete or partial response will undergo prophylactic cranial irradiation (PCI) within 1-30 days after completion of chemoradiotherapy, followed by adebrelimab monotherapy (1200 mg intravenously every 3 weeks) as consolidation and maintenance for up to 24 months in the absence of progression or unacceptable toxicity.

Treatment will be discontinued if the patient develops progressive disease, experiences unacceptable drug-related toxicity, withdraws consent, or meets any other pre-specified withdrawal criterion. Both efficacy (objective response rate, progression-free survival, overall survival) and safety (adverse events graded by CTCAE v5.0) endpoints will be assessed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years, either sex. Histologically or cytologically confirmed limited-stage small-cell lung cancer (LS-SCLC) defined by Veterans Administration Lung Group (VALG) two-stage system.

Availability of either an archival tumour-tissue block/slides or a newly obtained biopsy from a lesion that has not previously been irradiated.

≤ 2 prior cycles of chemotherapy or chemotherapy-naïve. ECOG performance-status 0 or 1. At least one measurable lesion per RECIST 1.1: ≥ 10 mm in longest diameter for non-nodal lesions or ≥ 15 mm in short axis for lymph-node lesions on CT scan.

Estimated life expectancy ≥ 3 months. Adequate pulmonary function (as judged by the investigator).

Adequate major organ function defined as:

Haematology: Hb ≥ 90 g/L; ANC ≥ 1.5 × 10⁹/L; PLT ≥ 100 × 10⁹/L. Biochemistry: serum albumin ≥ 30 g/L; ALT and AST < 3 × ULN; total bilirubin ≤ 1.5 × ULN; serum creatinine ≤ 1.5 × ULN.

Women of child-bearing potential must have a negative serum or urine pregnancy test within 14 days before enrolment and must use effective contraception from screening until ≥ 8 weeks after the last study-dose; men must be surgically sterile or agree to use effective contraception during the same period.

Voluntary informed consent signed; willing and able to comply with study procedures and follow-up.

Exclusion Criteria:

* Prior solid-organ, allogeneic stem-cell or planned transplantation. Immunosuppressive therapy ≤ 14 days before first adebrelimab dose (except intranasal/inhaled corticosteroids or physiological systemic doses equivalent to ≤ 10 mg/day prednisolone).

Known hypersensitivity to etoposide, cisplatin, adebrelimab, their excipients, or severe allergic reaction to any other monoclonal antibody.

Live-attenuated vaccine within 4 weeks before first dose or intent to receive one during the study.

Active autoimmune disease or history of autoimmune disease (e.g., autoimmune hepatitis, interstitial pneumonitis, uveitis, colitis, hypophysitis, vasculitis, nephritis, hyper-/hypothyroidism).

Uncontrolled asthma requiring bronchodilators or other systemic therapy (childhood asthma fully resolved and requiring no intervention in adulthood is allowed).

Urinalysis ≥ ++ protein or 24-h urine protein ≥ 1.0 g. Prior malignancy except adequately treated basal-cell or squamous-cell skin carcinoma or cervical carcinoma in situ.

HIV infection or known AIDS. Within 6 months before enrolment: myocardial infarction, severe/unstable angina, NYHA class ≥ II heart failure, poorly controlled arrhythmia (including QTcF > 450 ms [men] or > 470 ms [women] by Fridericia), symptomatic congestive heart failure.

Systemic anti-infective therapy (IV antibiotics, antifungals, or antivirals) within 4 weeks before first dose, or unexplained fever > 38.5 °C during screening or before first dose.

Active hepatitis B (HBV DNA ≥ 500 IU/mL), hepatitis C (anti-HCV positive and HCV-RNA detectable), or HBV/HCV co-infection.

Participation in another interventional clinical trial within 4 weeks before first dose.

Known history of substance abuse or recreational drug use. Any severe medical, psychiatric, or laboratory abnormality that, in the investigator's opinion, could increase study-related risk or interfere with results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-03-30 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
PFS | through study completion, an average of 3 years
  From subject enrollment to the first recorded disease progression or death from any cause, whichever occurs first

SECONDARY OUTCOMES:
ORR | through study completion, an average of 3 years
  The proportion of subjects achieving complete response (CR) or partial response (PR) as their best overall response following treatment initiation, relative to the total number of subjects.
OS | through study completion, an average of 3 years
  Time from subject enrollment to death from any cause.
DCR | through study completion, an average of 3 years
  The proportion of subjects achieving complete response (CR), partial response (PR), or stable disease (SD) as their best overall response following treatment initiation, relative to the total number of subjects.
Adverse Events | From the first dose of durvalumab to 90 days after the last dose of durvalumab or start of subsequent anticancer treatment
  AEs that occurred from the first dose of durvalumab to 90 days after the last dose of durvalumab or start of subsequent anticancer treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Cancer Hospital and Institute, Beijing, Beijing Municipality, China